CLINICAL TRIAL: NCT02568657
Title: Comparison Between Celox Versus Bakri Balloon for Treatment of Primary Atonic Postpartum Hemorrhage
Brief Title: Uterine Tamponade for Treatment of Primary Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Celox
Record Dates: First submitted 2015-10-04; First posted 2015-10-06 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celox group (Active Comparator): Celox placement is very simpe . During cesarean section celox is loaded in the lower uterine segment and part of it is passed through the cervix to the vagina. If PPH occurs after vaginal delivery the celox is inserted through the cervix to pack the lower uterine segment. Removal of Celox after 24 hours.
  Interventions: Device: Celox group
- Bakri balloon group (Active Comparator): Before insertion the balloon, ensure that the bladder is empty by placing a Foley catheter. Grasp the cervix with ring forceps. Insert the balloon into the cavity of the uterus under ultrasound guidance; making sure that the entire portion of the balloon passes the cervical canal above the internal cervical os. Once the correct placement is confirmed, inflate the balloon with sterile saline using the enclosed syringe.
  Interventions: Device: Bakri Balloon

INTERVENTIONS:
Device: Celox group
  Arms: Celox group
Device: Bakri Balloon
  Arms: Bakri balloon group

SUMMARY:
Postpartum hemorrhage (PPH) is responsible for around 25% of maternal mortality worldwide reaching as high as 60% in some countries.

Postpartum hemorrhage is defined as loss of 500 mL or more in a vaginal delivery and 1 Litre or more in a cesarean delivery.Also any blood loss that cause hemodynamic instability should be considered a PPH.

In 2012, WHO updated the guidelines for the management of PPH and retained placenta to include: "The use of intrauterine balloon tamponade is recommended for the treatment of PPH due to uterine atony. This recommendation is now stronger than the previous guidelines. It can be used for women who do not respond to uterotonics or if uterotonics are not available. This procedure potentially can avoid surgery and is appropriate while awaiting transfer to a higher-level facility".Furthermore, FIGO included Uterine balloon tamponade as a recommended second-line intervention for the treatment of PPH in their updated guidelines issued in 2012.

In 2006, the ACOG Practice Bulletin, published by the American College of Obstetricians and Gynecologists, made mention of the Bakri postpartum balloon for its specifically tailored design that enables conservative management of uterine bleeding in cases of uterine atony and other causes of PPH.

The reports demonstrated that balloon tamponade is helpful in managing PPH secondary to a wide variety of causes in resource-poor settings.

One of the new methods that could be used to control PPH is Uterine packing with chitosan-covered gauze or Celox.

Celox Haemostats are dressings with natural material called chitosan to control major haemorrhage including life-threatening bleeding . They are simple and effective, stopping major bleeding.It was first used by military forces to stop sever bleeding in the scene with no other options to stop bleeding. Celox™ granules are actually very high surface area flakes. When they come in contact with blood, Celox™ swells, gels, and sticks together to make a gel like clot, without generating any heat. Celox™ does not set off the normal clotting cascade, it only clots the blood it comes directly into contact with. Celox works on casualties using anticoagulants and anti-platelet therapy such as aspirin .

DETAILED DESCRIPTION:
Balloon tamponade is helpful in managing PPH secondary to a wide variety of causes in resource-poor settings.

One of the new methods that could be used to control PPH is Uterine packing with chitosan-covered gauze or Celox.

Celox Haemostats are dressings with natural material called chitosan to control major haemorrhage including life-threatening bleeding . They are simple and effective, stopping major bleeding.It was first used by military forces to stop sever bleeding in the scene with no other options to stop bleeding. Celox™ granules are actually very high surface area flakes. When they come in contact with blood, Celox™ swells, gels, and sticks together to make a gel like clot, without generating any heat. Celox™ does not set off the normal clotting cascade, it only clots the blood it comes directly into contact with. Celox works on casualties using anticoagulants and anti-platelet therapy such as aspirin.

We will be having two groups:

1. Celox group:

   Celox placement is very simpe . During cesarean section celox is loaded in the lower uterine segment and part of it is passed through the cervix to the vagina. If PPH occurs after vaginal delivery the celox is inserted through the cervix to pack the lower uterine segment. Removal of Celox after 24 hours.
2. Bakri balloon group:

Before insertion the balloon, ensure that the bladder is empty by placing a Foley catheter. Grasp the cervix with ring forceps. Insert the balloon into the cavity of the uterus under ultrasound guidance; making sure that the entire portion of the balloon passes the cervical canal above the internal cervical os. Once the correct placement is confirmed, inflate the balloon with sterile saline using the enclosed syringe.

ELIGIBILITY:
Inclusion Criteria:

1. Women who accept to participate (either the patient or her first-kin if she is unconscious)
2. Primary atonic postpartum hemorrhage

Exclusion Criteria:

1. Traumatic postpartum haemorrhage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss (mL) | 8 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374